CLINICAL TRIAL: NCT06733701
Title: The Use of Virtual Reality Technology During Oocyte Retrieval for in Vitro Fertilization: a Randomized Controlled Pilot Study
Brief Title: The Use of Virtual Reality Technology During Oocyte Retrieval for in Vitro Fertilization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Reproductive Endocrinology and Infertility (Unknown)
Responsible Party: Principal Investigator, Claire Jones, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-0033-E
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Oocyte Retrieval; Adverse Events; Procedural Anxiety; Pain Intensity; Satisfaction; Medication Administration
Keywords: Virtual Reality; Oocyte Retrieval; In Vitro Fertilization; Randomized Control Trial
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This will be a randomized, single-blinded, two-arm pilot study. Due to the nature of the intervention, participants cannot be blinded to allocation, but the physician performing the oocyte retrieval will be blinded to minimize the risk of bias.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): During the procedure, patients will receive standard of care analgesia and VR-based intervention (VRReliever Software V0.3.4 fromXRHealth)
  Interventions: Device: VR-based intervention (VRReliever Software V0.3.4 fromXRHealth)
- Control (Placebo Comparator): VR headset without any scenery
  Interventions: Device: VR headset without any scenery

INTERVENTIONS:
Device: VR-based intervention (VRReliever Software V0.3.4 fromXRHealth) — The participant will be able to select between four VR environments: beach, lake, forest, or mountain scenery. Each provides an immersive audio and visual environment designed to reduce anxiety and promote relaxation. Each scene is rendered in a high-resolution and life-like fashion which participants can experience in a full 360 degrees. Participants will wear the headset for the duration of the egg retrieval procedure which is approximately 15-20 minutes.
  Arms: Intervention
Device: VR headset without any scenery — VR headset without any scenery
  Arms: Control

SUMMARY:
Ultrasound-guided oocyte retrieval (OR) is a short, but oftentimes painful procedure, during which the follicles are punctured trans-vaginally to obtain oocytes for in vitro fertilization (IVF). Conscious sedation is the most commonly used method of pain relief, yet several studies have shown that more than half of women report moderate to high levels of pain and up to 7% of women report extreme or unacceptable levels of pain during OR. Adjuvant virtual reality (VR) therapy has been explored to reduce psychological stress during dental procedures, burn wound care, colonoscopy, as well as other minor procedures. Hence, the purpose of this study is to evaluate the use of VR technology during IVF treatment, particularly with respect to tolerability, patient satisfaction, and pain reduction during oocyte retrieval.

DETAILED DESCRIPTION:
Background / Rationale

Ultrasound-guided oocyte retrieval (OR) is a short, but oftentimes painful procedure, during which the follicles are punctured trans-vaginally to obtain oocytes for in vitro fertilization (IVF). Conscious sedation is the most commonly used method of pain relief, yet several studies have shown that more than half of women report moderate to high levels of pain and up to 7% of women report extreme or unacceptable levels of pain during OR. Psycho-social factors such as anxiety, previous negative experiences with gynecological examinations, and perceived lack of control are important predictors of OR-related pain. This finding is consistent with the multidimensionality of the pain experience. Although several adjuvant therapies have been proposed to reduce psychological stress during ART (assisted reproductive technology) therapy, their impact on the OR experience has been mixed.

Virtual reality (VR) allows users to engage in a fully immersive simulated environment using an advanced visual and auditory system. Multimodal stimuli contribute to a sense of actual presence/immersion in the virtual world, thus making the VR experience distinct from passive visual or auditory stimuli. The utility of VR therapy has been explored for numerous health applications, showing positive outcomes in clinical conditions such as dental procedures, burn wound care, colonoscopy, as well as other minor procedures. A recent systematic review of 39 RCTs (randomized clinical trials) concluded that VR's immersive, entertaining effects are useful for redirecting a patient's attention away from painful treatment experiences and reducing anxiety, discomfort, and unpleasantness. Several studies have shown a significant decrease in pain perception and anxiety scores when treated with VR, as measured by anxiety questionnaires, pulse rate reduction, and electroencephalogram changes compared with controls. To the best of our knowledge, there are no published studies that examine the application of VR technology during IVF treatment, particularly with respect to tolerability, patient satisfaction, and pain reduction during oocyte retrieval.

Purpose

The primary objectives of this pilot study are to evaluate patient acceptance, perceived utility, and adverse effects of VR technology during the oocyte retrieval procedure as measured by validated VR-engagement and anxiety-related questionnaires

ELIGIBILITY:
Inclusion Criteria:

- All adults undergoing their first oocyte retrieval

Exclusion Criteria:

* severe visual impairment
* contraindications to using VR technology according to manufacturer specifications including:
* severe motion sickness
* epilepsy/previous seizure
* claustrophobia
* current migraine
* heart disease
* use of medical devices such as cardiac pacemaker or hearing aids

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction and immersion | 10 minutes
  measured by the IGroup Presence Questionnaire (IPQ) -Scaled 14-item questionnaire administered post-OR
Adverse events | 20 minutes
  measured by the Simulator Sickness Questionnaire (SSQ) - Scaled 16-itemquestionnaire administered pre-OR and post-OR.
Procedural anxiety | 20 minutes
  measured by the State-Trait Anxiety Inventory (STAI) Questionnaire -Scaled 20-item questionnaire administered at recruitment, pre-OR, and post-OR.

SECONDARY OUTCOMES:
Pain intensity | 10 minutes
  using the Numerical Rating Scale (20)
Total opioid and benzodiazepine use | 20 minutes
  Dose for the procedure
Duration of procedure | 20 minutes
Total number of oocytes retrieved / peak E2 | 20 minutes
Total number of MII oocytes retrieved / number of follicles ≥ 17mm on day of trigger | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Claire Jones, MD, Principal Investigator — MOUNT SINAI HOSPITAL

IPD SHARING:
Plan to Share IPD: No
There are too few participants in the trial that they could potentially be identifiable.

REFERENCES:
- [Background] Frederiksen Y, Mehlsen MY, Matthiesen SM, Zachariae R, Ingerslev HJ. Predictors of pain during oocyte retrieval. J Psychosom Obstet Gynaecol. 2017 Mar;38(1):21-29. doi: 10.1080/0167482X.2016.1235558. Epub 2016 Sep 27. PMID 27670651
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Gejervall AL, Stener-Victorin E, Cerne A, Borg K, Bergh C. Pain aspects in oocyte aspiration for IVF. Reprod Biomed Online. 2007 Feb;14(2):184-90. doi: 10.1016/s1472-6483(10)60786-9. PMID 17298721
- [Background] Kwan I, Wang R, Pearce E, Bhattacharya S. Pain relief for women undergoing oocyte retrieval for assisted reproduction. Cochrane Database Syst Rev. 2018 May 15;5(5):CD004829. doi: 10.1002/14651858.CD004829.pub4. PMID 29761478